CLINICAL TRIAL: NCT05306639
Title: Effect of Spinal Magnetic Stimulation Versus Posterior Tibial Neuromodulation in Treatment of Monosymptomatic Nocturnal Enuresis: a Prospective Randomized Clinical Trial
Brief Title: Treatment of Monosymptomatic Nocturnal Enuresis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Nehad Mohamed Elshatby Mahmoud, Physician, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0305491
Record Dates: First submitted 2022-03-13; First posted 2022-04-01 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Nocturnal Enuresis
Keywords: spinal magnetic stimulation, nocturnal enuresis, neuromodulation
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal magnetic stimulation (Experimental): Spinal magnetic stimulation group will receive repetitive spinal magnetic stimulation sessions for a total of 12 sessions. Using the Neuro-MS/D machine, circular coil will be used to stimulate S2,3 and 4 sacral roots. The outer rim of the coil will be positioned in the midline over the sacral vertebrae (approximately 5 cm above the natal cleft, which approximates to the level of S2) Intensities will be adjusted to 50-70 % of maximal output (2.2 Tesla), stimulation frequency will be fixed at 15 Hz, burst length = 10 seconds, inter-burst interval = 30 seconds with a total of 1500 pulses
  Interventions: Other: Rehabilitation
- Neuromodulation (Experimental): Neuromodulation group will receive 12 sessions of bilateral transcutaneous posterior tibial neuromodulation using (Myomed 632®, Enraf Nonius, Delft, Netherlands) machine, the active rubber surface was placed behind the medial malleolus and the reference electrode was placed 10 cm proximal. Adjustment of the electric current was as follows: continuous current, pulse duration 200 ms, frequency 20 Hz; each session lasts for 30 min. The current intensity was adjusted according to the tolerance of the patient or until the big toe curls into plantar flexion
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — rehabilitation sessions using spinal magnetic stimulation or neuromodulation

SUMMARY:
A prospective randomized trial to study the effect of spinal magnetic stimulation versus posterior tibial neuromodulation in the treatment of monosymptomatic nocturnal enuresis.

DETAILED DESCRIPTION:
Nocturnal enuresis is defined as "nighttime bedwetting in children aged five years or older.Currently available treatment options for nocturnal enuresis include medication, wetting alarms, lifestyle changes, sacral magnetic stimulation, and posterior tibial neurmodulation.

Magnetic stimulation is a valid method for stimulation of sacral as functional electrical stimulation. It generates a more powerful and deeper electrical field than that produced by conventional electrical stimulators. So, magnetic stimulation could be considered an attractive form of electrical therapy, being relatively painless, non-invasive and free from side effects.Peripheral neuromodulation is the modulation of the physiologic behavior of the nerve by electrical stimulation. Posterior tibial neuromodulation is an effective method in treatment of urinary incontinence

ELIGIBILITY:
Inclusion Criteria:

* All subjects were diagnosed as patients with MNE according to the Diagnostic and statistical manual of mental disorders, 4th revised edition (DSM-IV) (American Psychiatric Association's DSM-IV, 1994): bed-wetting ≥3 times a week; lasting more than 6 months; can control urination during the day but cannot control urination after falling asleep.

Exclusion Criteria:

* - Patients younger than 5 years old.
* Patients who have any abnormality in blood or urine biochemistry.
* Patients with other urinary symptoms.
* Patients with neurological or endocrinal abnormalities (such as cerebral palsy, spinal cord lesion, peripheral neuropathy or diabetes mellitus)

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of bed wetting | one month
  Number of bed wettings/ week
Visual analogue scale to determine how much the enuresis affected his/her life. | three months
  Visual analogue scale from zero to ten (zero indicates no effect, 10 indicates severe bothersome

CONTACTS AND LOCATIONS:
Overall Officials: Nehad ElShatby, Principal Investigator — Alexandria University
Locations (1):
- Nehad ElShatby, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be available with the corresponding author to be shared with other researchers for three years after publishing the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: three years after publication
Access Criteria: Researchers can contact the corresponding author directly through e-mail